CLINICAL TRIAL: NCT03521986
Title: Postoperative Pain and Quality of Life for Patients Undergoing Mediastinal Tumor Resection by Subxiphoid and Intercostal VATS：A Randomized Controlled Trial
Brief Title: Pain and Quality of Life After Mediastinal Tumor Resection by Subxiphoid and Intercostal VATS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lei Jiang (Other)
Responsible Party: Sponsor-Investigator, Lei Jiang, Principal Investigator, Shanghai Pulmonary Hospital, Shanghai, China
Organization: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: leijiang2
Record Dates: First submitted 2018-04-30; First posted 2018-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Mediastinal Neoplasms; Thoracic Neoplasm; Thoracic Surgery
Keywords: Mediastinal Neoplasms; Pain; Quality of life
MeSH Terms: conditions — Mediastinal Neoplasms; Thoracic Neoplasms; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subxiphoid uniportal VATS (Experimental): Standard Subxiphoid single-port video assisted mediastinal thymectomy, no use of rib-spreader.
  Interventions: Procedure: Subxiphoid uniportal VATS
- Intercostal uniportal VATS (Active Comparator): Standard Intercostal single-port video assisted mediastinal thymectomy, no use of rib-spreader.
  Interventions: Procedure: Intercostal uniportal VATS

INTERVENTIONS:
Procedure: Subxiphoid uniportal VATS — Patients were placed in a supine position, and the operating table was manipulated as needed to elevate the appropriate side of the body for surgery. The surgical procedures followed principles of pulmonary resections
  Arms: Subxiphoid uniportal VATS
Procedure: Intercostal uniportal VATS — The surgical procedures followed principles of pulmonary resections
  Arms: Intercostal uniportal VATS

SUMMARY:
Thoracoscopic assisted mediastinal thymectomy is currently one of the most commonly used surgical methods, but there are some deficiencies.Minimally invasive surgery through the subxiphoid approach can achieve a good surgical field of vision. (1) The surgical field is fully exposed. (2) damage to intercostal nerves can be avoided.(3) Operation time, intraoperative blood loss, postoperative Extubation time is similar to VATS. But there is still lack of evidence.

In this study, 50 patients undergoing subxiphoid uniportal VATS and 50 patients undergoing intercostal uniportal VATS were included to evaluate the post-operative pain and quality of life after surgery.

DETAILED DESCRIPTION:
The types of tumors in the medial mediastinal area were different. Thymoma, germ cell tumors, ectopic parathyroid tumors, and lymphoid tumors were in the anterior mediastinum. Bronchial cysts, pericardial cysts, and lymphomas were in the middle mediastinum. The principles of treatment for mediastinal tumor surgery must be both safe and radical. Radical resection is the dominant position in the treatment of mediastinal tumors, including traditional open surgery and thoracoscopic assisted minimally invasive surgery. At present, minimally invasive surgery for mediastinal tumor includes video-assisted thoracoscopic surgery via subxiphoid approach, left or right intercostal approach, trans-cervical approach and "Da Vinci" robotic system. Compared with conventional sternotomy, thoracoscopic assisted minimally invasive mediastinal tumor resection has clearer, multi-angle surgical vision, less trauma, less intraoperative blood loss, early postoperative extubation, and short postoperative hospital stay, postoperative recovery faster, less pain, fewer complications and meet the beauty needs and so on. Thoracoscopic assisted mediastinal thymectomy is currently one of the most commonly used surgical methods, but there are some deficiencies.

Minimally invasive surgery through the subxiphoid approach can achieve a good surgical field of vision. Compared with the traditional transcostal VATS medial mediastinal tumor resection, the subxiphoid thoracoscopic surgery had obvious advantages: (1) The surgical field is fully exposed. For patients with myasthenia gravis, it is particularly necessary to clean bilateral mediastinal adipose tissue; (2) Without intercostal surgery, damage to intercostal nerves can be avoided, postoperative pain can be reduced, and quality of life can be improved; (3) Operation time, intraoperative blood loss, postoperative Extubation time is similar to VATS. Disadvantages are as follows: (1) If there is a large hemorrhage during surgery, an emergency transfer to open the chest is required. The injury is greater and the operation is more troublesome; (2) Anterior septal space is Smaller, surgical instruments are more likely to interfere with each other. But there is still lack of evidence to prove which is better.

In this study, 100 patients with anterial and middle mediastinal tumors were selected as study subjects. 50 patients undergoing subxiphoid uniportal VATS were included in the observation group, and 50 patients undergoing intercostal uniportal VATS were included in the control group. The operation time, incision length, intraoperative blood loss, postoperative drainage time, postoperative drainage, hospitalization and hospitalization costs of the 2 groups would be observed. The clinical efficacy and incidence of complications were compared between the 2 groups. After six months of follow-up, postoperative pain and postoperative quality of life were observed in the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of anterial and middle mediastinal tumors ;
2. Normal heart function, pulmonary function FEV1 %> 60% PaO2> 80 mmHg
3. BMI<30

Exclusion Criteria:

1. enlargement of lymph nodes was seen in the clinical CT readings.
2. Preoperative chronic pain or chronic opioid analgesics
3. Preoperative check for mental disorders such as hyper-anxiety
4. History of previous thoracic surgery
5. Patients with thoracic deformity (eg, funnel chest and chicken breast)
6. Poor education can not understand postoperative follow-up requirements and assessment scale

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-04-04 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | 6 months
  visual analogue score (VAS-score) is to asses the development of acute and chronic pain after VATS surgery. 11 point numeric rating scale of 0 represented "no pain"and a score of 10 represented "worst pain ".

SECONDARY OUTCOMES:
Quality of life | 6 months
  the EuroQol 5 Dimensions (EQ5D) and European Organisation for Research and Treatment of Cancer (EORTC) 30 item Quality of Life Questionnaire (QLQ-C30) are used. EQ5D includes self-reported quality of life, where 0 is the worst and 100 is the best imaginable health state. QLQ-C30 is a 30-item questionnaire, from which six functional domains of quality of life (physical function, emotional function, cognitive function, social function, and role function), and nine symptom domains (fatigue, pain, nausea and vomiting, dyspnoea, insomnia, appetite, constipation, diarrhoea, and financial difficulties) can be extracted, as well as an overall score.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes